CLINICAL TRIAL: NCT04091971
Title: Examining the Effects of Ketamine Treatment on Synaptic Plasticity in Depression Using PET Imaging
Brief Title: Ketamine Treatment Effects on Synaptic Plasticity in Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Jeffrey Miller, Director of Brain Imaging, Division of Molecular Imaging and Neuropathology, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7847
Record Dates: First submitted 2019-09-11; First posted 2019-09-17 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Depressed adults with current major depressive disorder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Depressed adults with current MDD (Experimental): Subjects will undergo 4 sequential intravenous infusions of ketamine administered over a two week period.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Subjects will undergo 4 sequential intravenous infusions of ketamine administered over a two week period.
  Ketamine is administered at a dose of 0.5mg/kg intravenously as a slow continuous infusion over approximately 40 minutes, with 4 sequential infusions over an approximately two week period (two infusions per week for two weeks).

SUMMARY:
Depression is the leading cause of disability globally (1, 2). One-third to one-half of patients suffering from major depressive disorder (MDD) do not achieve remission even after multiple antidepressant trials (3). Ketamine is a commonly-used FDA-approved anesthetic medication that at subanesthetic doses leads to rapid antidepressant and anti-suicidal ideation effects in hours, rather than weeks, following administration. Despite these promising findings, a key limitation of ketamine treatment is that it only yields an antidepressant response in approximately 50% of those treated. The goal of this project is to A) elucidate ketamine's mechanism of action and B) identify biomarkers predicting treatment outcome to ketamine which could be used to match patients to treatment based on the likelihood of effectiveness at the individual level. Data from animal models suggests that ketamine acts by enhancing the connections between neurons through a process known as synaptic plasticity (4-7), and that these biological changes are responsible for the sustained behavioral effects of ketamine (8). A newly available tool allows us to image the density of these synaptic connections in the living brain using PET (positron emission tomography) imaging with a radiotracer called [11C]UCB-J, which is a marker of synaptic density. We propose to directly quantify synaptic density in depressed patients before and after a course of ketamine, to examine changes in density following treatment. In exploratory analyses, we will examine synaptic density as a mediator of the sustained antidepressant effects of ketamine and as a predictor of treatment outcome. To study these questions, we will quantify synaptic density using PET imaging before and after a course of 4 sequential intravenous infusions of ketamine administered over a two week period. Study participation involves an inpatient stay of approximately three weeks at the New York State Psychiatric Institute at no cost.

DETAILED DESCRIPTION:
Depression is the leading cause of disability globally (1, 2). One-third to one-half of patients suffering from major depressive disorder (MDD) do not achieve remission even after multiple antidepressant trials (3). Ketamine is a commonly-used FDA-approved anesthetic and non-competitive N-methyl-D-aspartate (NMDA) glutamate receptor antagonist. Recent randomized trials demonstrate that subanesthetic doses of ketamine lead to rapid antidepressant and antisuicidal ideation effects in individuals with MDD and bipolar depression (reviewed in (9)). In contrast to current FDA-approved antidepressants, ketamine exerts antidepressant effects in hours, rather than weeks, following administration. Despite these promising findings, a key limitation of ketamine treatment is that it only yields an antidepressant response in approximately 50% of those treated. In addition, ketamine's clinical utility is limited by its acute dissociative side effects, a one to two-week duration of action as monotherapy, its addictive potential, and long term safety concerns related to cognition and interstitial cystitis (9-11). Given the profound benefit of ketamine for some individuals yet these key limitations, developing a precision medicine research strategy for ketamine's antidepressant effects could be of tremendous scientific and clinical benefit, in order to A) elucidate ketamine's mechanism of action, to advance the development of safer alternative agents and B) identify biomarkers predicting treatment outcome to ketamine, which could be used to match patients to treatment based on the likelihood of effectiveness at the individual level.

There is evidence of brain atrophy in depression: gray matter volume is reduced in the prefrontal cortex (PFC) and in the hippocampus (HC) in depressed individuals (12). Postmortem studies in depression show low expression of several genes related to synaptic function and decreased synapse number in the dorsolateral PFC (13). Chronic stress, a risk factor for depression, precipitates neuronal atrophy and dendritic spine loss in HC and PFC (14, 15). Preclinical work in rodents suggests that ketamine may exert antidepressant effects by reversing neuronal atrophy, specifically through the formation of new dendritic spine synapses in the brain. In rodents, ketamine induces rapid synaptogenesis via stimulation of mechanistic target of rapamycin (mTOR) and brain-derived neurotrophic factor (BDNF), leading to a reversal of chronic, stress-induced neuronal atrophy (4-7).

A recently developed research tool enables examination of synaptic density in vivo in humans. [11C]UCB-J is a PET radiotracer that is specific for synaptic vesicle glycoprotein 2A (SV2A) (16, 17), providing a quantitative measure of synaptic density in vivo in the brain in humans. A recent PET imaging pilot study identified low [11C]UCB-J binding in the PFC of individuals with current MDD as compared to healthy volunteers, providing early evidence that this synaptic density biomarker may quantify a disease-relevant process in depression (18). Furthermore, PET imaging with [11C]UCB-J displays outstanding test-retest reliability, with absolute test-retest variability of only 4-5% in brain regions of interest in this study (19), making it an outstanding tool for longitudinal studies of the effects of treatment interventions. We therefore propose to directly quantify synaptic density in depressed patients to investigate whether it is increased by treatment with ketamine in a regionally-specific manner. Moreover, we will examine synaptic density as a mediator of the sustained antidepressant effects of ketamine and as a predictor of treatment outcome. We will quantify synaptic density using PET imaging before and after a course of 4 sequential intravenous infusions of ketamine administered over a two-week period. Study participation involves an inpatient stay of approximately three weeks at the New York State Psychiatric Institute at no cost.

ELIGIBILITY:
Inclusion Criteria:

* Unipolar, major depressive episode (MDE), with 17-item Hamilton Depression Rating Scale score ≥16. Patients may be psychiatric medication- free, or if currently taking psychiatric medication, not responding adequately as evidenced by current MDE.
* 18-55 years old
* Female patients of child-bearing potential must be willing to use an acceptable form of birth control during study participation such as condoms, diaphragm, oral contraceptive pills.
* Must be enrolled in division's umbrella research protocol
* Able to provide informed consent
* Agrees to voluntary admission to an inpatient research unit at The New York State Psychiatric Institute (NYSPI) for baseline PET imaging and Magnetic Resonance Imaging (MRI), ketamine infusion, and repeat PET imaging

Exclusion Criteria:

* Unstable medical or neurological illness including: A) baseline hypertension (BP>140/90); B) significant history of cardiovascular illness; C) Platelet count < 80,000 cells/uL; and D) Hemoglobin < 11 g/dL for females and < 12 g/dL for males
* Significant electrocardiogram (ECG) abnormality (e.g., Ventricular tachycardia, evidence of myocardial ischemia, symptomatic bradycardia, unstable tachycardia, second degree (or greater) atrioventricular (AV) block).
* Pregnancy, currently lactating, or planning to conceive during the course of study participation.
* Diagnosis of bipolar disorder or current psychotic symptoms.
* Current or past ketamine use disorder (lifetime); any drug or alcohol use disorder within past 6 months
* Inadequate understanding of English.
* Prior ineffective trial of or adverse reaction to ketamine.
* A neurological disease or prior head trauma with evidence of cognitive impairment.

Subjects who endorse a history of prior head trauma and score ≥ 1.5 standard deviations below the mean on the Trailmaking A&B will be excluded from study participation.

- Metal implants or paramagnetic objects contained within the body (including heart pacemaker, shrapnel, or surgical prostheses) which may present a risk to the subject or interfere with the MRI scan, according to the guidelines set forth in the following reference book commonly used by neuroradiologists: "Guide to MR procedures and metallic objects," F.G. Shellock, Lippincott Williams and Wilkins NY 2001. Additionally transdermal patches will be removed during the MR study at the discretion of the investigator.

* Current, past, or anticipated exposure to radiation, that may include: **
* being badged for radiation exposure in the workplace
* participation in nuclear medicine research protocols in the last year
* Claustrophobia significant enough to interfere with MRI scanning
* Weight that exceeds 325 lbs or inability to fit into MRI scanner
* Individuals taking prescribed opioid medication, using opioids recreationally, or taking naltrexone at the time of enrollment 14. Daily use of: benzodiazepine, zolpidem (Ambien), zaleplon (Sonata), or eszopiclone (Lunesta) for ≥2 weeks at time of consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute/Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
If a subject consents to participate in this research, their personal information will be kept confidential and will not be released without their written permission except as described in this section or as required by law. Data collected in this research study, including MRI and PET scans, measurements from blood samples drawn during the PET scan, and questionnaire answers, may be used in future studies, and may be shared with other investigators after being de-identified, including in scientific data banks. This means that information that identifies these data with their identity will be removed beforehand any data is shared. While the measurements we record from blood samples may be shared with other investigators after being de-identified, no biospecimens from this research study will be shared with other investigators.

RESULTS

PARTICIPANT FLOW:
Groups:
- Depressed Adults With Current MDD: Subjects will undergo 4 sequential intravenous infusions of ketamine administered over a two week period.
  Ketamine is administered at a dose of 0.5mg/kg intravenously as a slow continuous infusion over approximately 40 minutes, with 4 sequential infusions over an approximately two week period (two infusions per week for two weeks).
Period: Overall Study
Arm/Group | Depressed Adults With Current MDD
Started | 9
Completed | 5
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — No longer met eligibility criteria after enrollment. | 2
Not completed — Panic attack during MRI; no MRI or PET but completed ketamine and other procedures | 1

BASELINE CHARACTERISTICS:
Population: Including only participants who completed research procedures beyond initial screening and consent (n=6: 5 completers and 1 participants with clinical outcomes but not PET)
Groups:
- Depressed Adults With Current MDD: Subjects will undergo 4 sequential intravenous infusions of ketamine administered over a two week period.
  Ketamine: See arm description.
Arm/Group | Depressed Adults With Current MDD
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.33 (3.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Synaptic Density
Description: PET imaging measure of synaptic density ([11C]UCB-J binding potential, BPND) before and after ketamine treatment. This type of brain scan takes pictures to measure the density of synapses, or connections between brain cells (neurons), in the brain. [11C]UCB-J is a radiotracer specific for SV2A, a protein present in presynaptic vesicles. [11C]UCB-J BPND was quantified in a brain region called the medial prefrontal cortex; previous studies have found lower levels of [11C]UCB-J binding in patients with more severe depression. BPND is the ratio at equilibrium of specifically bound radioligand to that of nondisplaceable radioligand in tissue.
  Time frame of assessment: Time frame 1 = baseline. This pre-treatment PET scan was acquired as close as possible prior to the first ketamine infusion, up to 7 days prior to first ketamine infusion. Time frame 2 = post-treatment. This post-treatment PET scan was acquired 24-48 hours following the final (4th) ketamine infusion.
Time Frame: Measured at two time frames: Time frame 1 = Baseline. Time frame 2 = post-treatment
Population: Participants with MDD who completed PET imaging pre-post a course of ketamine infusions for depression
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Depressed Adults With Current MDD
Number analyzed (Participants) | 5
Ratio
  Pre-treatment [11C]UCB-J binding potential (BPnd) in medial prefrontal cortex | 2.40 (0.81)
  Post-treatment [11C]UCB-J binding potential (BPnd) in medial prefrontal cortex | 2.32 (0.67)

2. Secondary Outcome: 17-item Hamilton Depression Rating Scale
Description: The 17-item Hamilton Depression Rating Scale (HDRS) is a clinician-administered scale that quantifies depression severity, and includes items assessing mood, suicidal thinking, insomnia, feelings of guilt, work and activities, somatic symptoms, and insight. It is a well-characterized scale with excellent psychometric properties. The version of the scale used in this study has a range from 0 to 51. Interpretation of score values is as follows:
  None: 0-7 Mild: 8-13 Moderate: 14-19 Severe: 20-25 Very Severe: 26-51
Time Frame: Measured at 3 time frames. Time frame one = Baseline: 24 hours prior to infusion one ("PRE"). Time frame two = 24 hours following ketamine infusion 4 ("POST1"). Time frame three = one week following ketamine infusion 4 ("POST2").
Population: Including all participants with HDRS data, n=6. 1 of the 6 does not have PET data. Including data from the 3 time points relevant for analysis: 24 hours prior to first ketamine infusion ("PRE"), 24 hours following ketamine infusion 4 ("POST1") and 1 week following ketamine infusion 4 ("POST2").
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Depressed Adults With Current MDD
Number analyzed (Participants) | 6
score on a scale
  HAM-17 24 hours prior to first ketamine infusion ("PRE") | 19.5 (3.0)
  HAM-17 24 hours following ketamine infusion 4 ("POST1") | 6.5 (2.4)
  HAM-17 1 week following ketamine infusion 4 ("POST2") | 7.8 (4.4)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: No differences
Groups:
- Depressed Adults With Current MDD: Subjects will undergo 4 sequential intravenous infusions of ketamine administered over a two week period.
  Ketamine: Ketamine is administered at a dose of 0.5mg/kg intravenously as a slow continuous infusion over approximately 40 minutes, with 4 sequential infusions over an approximately two week period (two infusions per week for two weeks).
Arm/Group | Depressed Adults With Current MDD
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Depressed Adults With Current MDD (N=9)
Insomnia (Nervous system disorders) | 2 (2) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Nightmares (Nervous system disorders) | 1 (1) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Drowsiness (Nervous system disorders) | 2 (4) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Feeling nervous or hyper (Nervous system disorders) | 1 (1) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Irritability (Nervous system disorders) | 2 (2) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Memory difficulties (Nervous system disorders) | 2 (7) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Trouble concentrating (Nervous system disorders) | 1 (1) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Headache (Nervous system disorders) | 2 (3) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Ringing in Ears or Trouble Hearing (Ear and labyrinth disorders) | 2 (2) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Drooling or Increased Salivation (General disorders) | 1 (1) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Heartbeat rapid or pounding (Cardiac disorders) | 1 (1) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Trouble catching breath or hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Chest pain (Cardiac disorders) | 1 (1) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Nausea or vomiting (Gastrointestinal disorders) | 1 (1) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Frequent need to urinate (Renal and urinary disorders) | 2 (4) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Loss of Sexual Interest (Reproductive system and breast disorders) | 1 (1) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Delayed or absent orgasm (Reproductive system and breast disorders) | 1 (5) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Excessive Sweating (General disorders) | 3 (6) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Decreased appetite (Gastrointestinal disorders) | 3 (4) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Increased appetite (Gastrointestinal disorders) | 1 (4) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Weight loss (General disorders) | 1 (2)
Skin rash or allergy (Skin and subcutaneous tissue disorders) | 1 (1) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Word finding difficulties (Nervous system disorders) | 1 (1) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Apathy/emotional indifference (Nervous system disorders) | 1 (1) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.
Hair thinning/loss (General disorders) | 2 (2) — Assessed by SAFTEE self-report at 8 time points after commencing ketamine. All items endorsed that were not present at at least the same level pre-ketamine assessed via SAFTEE are included in this table, whether related to study procedures or not.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT04091971/Prot_SAP_003.pdf